CLINICAL TRIAL: NCT04955678
Title: ZG-801 Phase III Trial - Randomized, Double-blind, Placebo-controlled Trial of ZG-801 in Patients With Hyperkalemia -
Brief Title: A Comparative Study of ZG-801 and Placebo in Patients With Hyperkalemia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Zeria Pharmaceutical (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ZG-801-02
Record Dates: First submitted 2021-07-01; First posted 2021-07-09 (Actual); Last update posted 2023-04-20 (Actual); Status verified 2022-10

CONDITIONS: Hyperkalemia
MeSH Terms: conditions — Hyperkalemia | interventions — Calcium

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ZG-801 (Experimental)
  Interventions: Drug: Calcium, hydrolysed divinylbenzene-Me 2-fluoro-2-propenoate-1, 7-octadiene polymer sorbitol complexes
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Calcium, hydrolysed divinylbenzene-Me 2-fluoro-2-propenoate-1, 7-octadiene polymer sorbitol complexes — ZG-801 is powder for suspension. In Run-in period, ZG-801 is taken once a day for 4 or 5 weeks. In Double-blind period, ZG-801 is taken once a day for 4 weeks.
  Arms: ZG-801
Drug: Placebo — Placebo is powder for suspension. In Double-blind period, Placebo is taken once a day for 4 weeks.
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the superiority of ZG-801 to placebo in Japanese hyperkalemia patients whose serum potassium value becomes normal in the Run-in period by comparing the change in the value at the Double-blind period week 4, and to further evaluate the efficacy and safety of ZG-801 in Japanese hyperkalemia patients administrated ZG-801 for maximum 9 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Patients whose serum potassium value (local) at the Run-in period baseline is ≥5.5mEq/L, < 6.5 mEq/L
* Age 20 - 80 years old at informed consent
* Patients who understand an overview of the study and voluntarily consented to participate in the study by documents.

Main Exclusion Criteria:

* Patients determined to require emergency treatment for hyperkalemia at the Run-in period baseline
* Patients with poorly controlled blood pressure
* Patients with heart failure in New York Heart Association Class IV
* Patients who have experienced heart transplant, liver transplant or kidney transplant or who are predicted that the need for them will occur during the study
* Patients who have taken any of the following medication within 7 days prior to the Run-in period baseline or currently administrated.

  1. Sodium polystyrene sulfonate
  2. Calcium polystyrene sulfonate
  3. Sodium zirconium cyclosilicate hydrate
  4. Potassium supplement
* Patients with or who have experienced a severe swallowing disorder, moderate to severe gastroparesis, severe constipation, bowel obstruction, incarceration, abnormal post-operative bowel motility disorders or severe gastrointestinal disorders. In addition, patients who have experienced bariatric surgery or major gastrointestinal surgery (e.g., bowel resection).
* Patients suspected to be with transient high potassium value.(ex. caused by dietary effects only)

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 85 (Actual)
Dates: Start 2021-08-03 (Actual); Primary Completion 2022-12-26 (Actual); Study Completion 2023-03-13 (Actual)

PRIMARY OUTCOMES:
Change in serum potassium value at Double-blind period week4 | Double-blind period baseline to Double-blind period week4

SECONDARY OUTCOMES:
Maintenance of serum potassium value within 3.5 mEq/L to < 5.1 mEq/L or within 3.5 mEq/L to <5.5 mEq/L in Double-blind Period | Double-blind period baseline to Double-blind period week4
Time to First Non-maintenance of Serum Potassium Value in Double-blind Period | Double-blind period baseline to Double-blind period week4
RAASi dose sustaining proportion | Double-blind period baseline to Double-blind period week4
Change in Serum Potassium Value | Run-in period baseline to Run-in period week 5

CONTACTS AND LOCATIONS:
Overall Officials: Yusuke Tomioka, Study Director — Zeria Pharmaceutical
Locations (1):
- Zeria Investigative Site, Hitachi-Naka, Ibaraki, Japan